CLINICAL TRIAL: NCT02927483
Title: A Comparative Study to Assess the Efficacy and Safety of Endolex Forte vs Diosmin and Hesperidin in Reducing the symptomatoLogy of Patients With ChronIc VeNous Insufficiency Between Functional Classes CEAP 1-4, During a Period of 6 Months
Brief Title: Study to Assess the Efficacy and Safety of Endolex Forte VErsus Diosmin and Hesperidin in Reducing VeNous Insufficiency
Acronym: EVELINE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SunWave Pharma (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPSUN/0116/FS
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Venous Insufficiency
Keywords: Venous Insufficiency
MeSH Terms: conditions — Venous Insufficiency | interventions — Hesperidin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endolex Forte® (Experimental): Endolex Forte® oral capsules administered from Baseline Visit until Day 180, two capsules per day.
  Interventions: Dietary Supplement: Endolex Forte®
- A combination of diosmin and hesperidin (Active Comparator): A combination of diosmin and hesperidin is a combination of micronized diosmin (450 mg) and micronized hesperidin (50 mg) film-coated tablets administered from Baseline Visit until Day 180, two tablets per day.
  Interventions: Dietary Supplement: A combination of diosmin and hesperidin

INTERVENTIONS:
Dietary Supplement: Endolex Forte® — Endolex Forte® oral capsules administered from Baseline Visit until Day 180, two capsules per day.
  Arms: Endolex Forte®
Dietary Supplement: A combination of diosmin and hesperidin — A combination of diosmin and hesperidin is a combination of micronized diosmin (450 mg) and micronized hesperidin (50 mg) film-coated tablets administered from Baseline Visit until Day 180, two tablets per day.
  Arms: A combination of diosmin and hesperidin

SUMMARY:
The trial is designed as a randomized, multicenter, open label, comparative, 6 months, clinical study.

DETAILED DESCRIPTION:
A randomized, multicentered, open label, comparative study to assess the efficacy and safety of Endolex Forte® versus a combination of micronized diosmin (450 mg) and micronized hesperidin (50 mg) in reducing the symptomatology of patients diagnosed with Chronic Venous Insufficiency which is rated between functional classes CEAP 1-4, during a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or females aged 18 to 75 years old
* BMI≤40
* Presence of chronic venous insufficiency which is rated between functional classes CEAP 1-4
* Patients diagnosed with superficial vein thrombophlebitis and have skin reaction by redness, swelling, fever and pain symptoms.or patients presenting a painful venous symptomatology in the lower limbs for at least 30 days.
* Willing and able to give written informed consent prior to participation in the trial
* Patients expected to be compliant with the study treatment

Exclusion Criteria:

* Known allergy to the product's ingredients
* Pregnancy or breastfeeding
* Patient is involved in any other clinical trial
* Deep vein thrombosis
* Stasis dermatitis
* The patient is taking non-steroids anti-inflammatory drugs include oral , topical creams or patch form)
* Open ulcers or lower extremity amputation
* Patient treated by venotonic treatments or vascular protectants or assimilated dietary supplements or homeopathic treatments or diuretics within 15 days prior inclusion
* Patient presenting permanent oedema,
* Patient with a history of lower limbs trauma responsible for sequel pains
* NYHA III and IV Heart Failure
* Renal Failure
* Untreated or uncontrolled Arterial Hypertension
* Hepatic Failure
* History of a known liver disease such as hepatitis A, hepatitis B, or C.
* Malignant neoplasms, from any etiology, or who are receiving any type of anticancer treatment, unless when properly treated and with no evidence of recurrence during the last five years
* Previous history of alcoholism, drug abuse, psychological or emotional problems in the last 5 years that can invalidate the Informed Consent Form or restrain participant's ability to comply with the requirements of the protocol.
* Immobility.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in limb volume determination at day 180 (water displacement method) | 180 days

SECONDARY OUTCOMES:
Change from baseline in limb volume determination at day 90 (water displacement method) | 90 days
Change from pre-treatment (baseline) in the calf circumference on treatment day 30 | 30 days
Change from pre-treatment (baseline) in the calf circumference on treatment day 180 | 180 days
Change from baseline in the subjective symptoms of CVI (tired, heavy legs, sensation of tension in the legs, pain in the legs) measured by Visual Analogue Scales (VAS) at day 90 | 90 days
Change from baseline in the subjective symptoms of CVI (tired, heavy legs, sensation of tension in the legs, pain in the legs) measured by Visual Analogue Scales (VAS) at day 180 | 180 days
Global assessment of efficacy by the investigator at day 180 | 180 days
Questionnaire on improvement in symptoms at day 180 (CIVIQ-20) | 180 days
Global assessment of tolerability by the investigator at day 180 | 180 days
Adverse events | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Calin Giurcaneanu, MD, Principal Investigator — Spitalul Universitar de Urgenta Elias, Sectia Dermatologie

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Eberhardt RT, Raffetto JD. Chronic venous insufficiency. Circulation. 2005 May 10;111(18):2398-409. doi: 10.1161/01.CIR.0000164199.72440.08. No abstract available. PMID 15883226
- [Background] Olin JW, Beusterien KM, Childs MB, Seavey C, McHugh L, Griffiths RI. Medical costs of treating venous stasis ulcers: evidence from a retrospective cohort study. Vasc Med. 1999;4(1):1-7. doi: 10.1177/1358836X9900400101. PMID 10355863
- [Background] Porter JM, Moneta GL. Reporting standards in venous disease: an update. International Consensus Committee on Chronic Venous Disease. J Vasc Surg. 1995 Apr;21(4):635-45. doi: 10.1016/s0741-5214(95)70195-8. PMID 7707568
- [Background] Rabe E, Stucker M, Ottillinger B. Water displacement leg volumetry in clinical studies--a discussion of error sources. BMC Med Res Methodol. 2010 Jan 13;10:5. doi: 10.1186/1471-2288-10-5. PMID 20070899
- [Background] Perrin M, Ramelet AA. Pharmacological treatment of primary chronic venous disease: rationale, results and unanswered questions. Eur J Vasc Endovasc Surg. 2011 Jan;41(1):117-25. doi: 10.1016/j.ejvs.2010.09.025. Epub 2010 Dec 3. PMID 21126890
- [Background] Monograph. Diosmin. Altern Med Rev. 2004 Sep;9(3):308-11. No abstract available. PMID 15387721
- [Background] Sezer A, Usta U, Kocak Z, Yagci MA. The effect of a flavonoid fractions diosmin + hesperidin on radiation-induced acute proctitis in a rat model. J Cancer Res Ther. 2011 Apr-Jun;7(2):152-6. doi: 10.4103/0973-1482.82927. PMID 21768702